CLINICAL TRIAL: NCT05359627
Title: A Pharmacokinetic Study of Polymyxin B in Healthy Subjects and Subjects With Renal Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TTYPX2201
Record Dates: First submitted 2022-03-29; First posted 2022-05-04 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Antibiotic Toxicity
MeSH Terms: interventions — Polymyxin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): normal renal function group
  Interventions: Drug: Polymyxin B
- Arm 2 (Experimental): mild renal insufficiency group
  Interventions: Drug: Polymyxin B
- Arm 3 (Experimental): long-term IHD group
  Interventions: Drug: Polymyxin B

INTERVENTIONS:
Drug: Polymyxin B — Polymyxin B acts against gram-negative bacteria (GNB) only, via three known mechanisms of action: First, polymyxin B can electrostatically interact with the outer membranes of GNB to compete against and displace calcium and magnesium divalent cations from membrane lipids, thereby disrupting lipopolysaccharide (LPS) molecules on the outer membrane and triggering their release. This leads to changes in the permeability of the bacterial membrane and subsequently causes cell content leakage, cell lysis, and death. Second, polymyxin B can act as a surfactant, as it is amphipathic and contains both lipophilic and lipophobic groups; this allows it to penetrate cell membranes, interact with the phospholipids within, and rapidly disrupt membranes to kill bacteria. Third, polymyxin B can bind to the lipid A portion of bacterial endotoxin or LPS molecules, thus neutralizing their toxicity.

SUMMARY:
This is an open-label, single-center, single-dose, parallel-group study to evaluate the PK and safety profiles of polymyxin B administered by IV infusion in healthy subjects and subjects with renal insufficiency.

DETAILED DESCRIPTION:
The study will enroll approximately 24 adult subjects in the following three Arms based on renal function. Approximately 8 subjects for each Arm are planned to be enrolled to fulfill the analysis of at least 6 evaluable subjects in each Arm. The subject who drops out of the study may be replaced at the discretion of the Sponsor.

* Arm 1 (normal renal function group): Subjects with CLcr ≥ 90 mL/min
* Arm 2 (mild renal insufficiency group): Subjects with CLcr between 60 and 89 mL/min (inclusive)
* Arm 3 (long-term IHD group): Subjects with ESRD receiving IHD therapy 3 times a week for at least 3 months prior to dosing of study drug; Subjects will receive a single dose of polymyxin B one day after his/her 3rd dialysis of the week.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 20 and 70 years of age (inclusive) at screening.
* Subjects with Body Mass Index (BMI) between 18.5 and 35 kg/m² (inclusive) at screening.
* Subjects with sitting heart rate between 60 and 100 beats/min at screening.
* Subjects with serum albumin between 3.5 and 5.7 g/dL (inclusive).
* Subjects (normal renal function group) with creatinine clearance (CLcr) ≥ 90 mL/min at screening; Subjects (mild renal insufficiency group) with CLcr between 60 and 89 mL/min (inclusive) within 3 months prior to screening and at screening; Subjects (long-term IHD group) with ESRD receiving IHD therapy 3 times a week for at least 3 months prior to dosing of study drug.
* Female subjects with childbearing potential must have a negative serum pregnancy test at screening and pregnancy test on Day -1.
* Subjects with sufficient peripheral vascular access for blood collection.
* Subject is willing and able to comply with all study procedures and restrictions.
* Subject understands the study procedures and is willing and able to provide written informed consent.

Exclusion Criteria:

* Arm 1 (normal renal function group): Subject with history or presence of any clinically significant cardiovascular, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, psychiatric disease or disorder, with active bleeding or with head injury or meningitis 3 months prior to dosing, in the opinion of the investigator or any uncontrolled medical illness which in the opinion of the investigator would jeopardize the safety of the subject, interfere with study assessments, or impact the validity of the study results; Arm 2 (mild renal insufficiency group): Subject with history or presence of any clinically significant cardiovascular, respiratory, hepatic, hematological, immunologic, neurological, psychiatric disease, active bleeding within 3 months, congenital renal disease (e.g., polycystic kidney disease) or disorder, with head injury or meningitis 3 months prior to dosing, in the opinion of the investigator or any uncontrolled medical illness which in the opinion of the investigator would jeopardize the safety of the subject, interfere with study assessments, or impact the validity of the study results; Arm 3 (long-term IHD group): Subject with history or presence of any clinically significant respiratory, hepatic, hematological, immunologic, neurological, psychiatric disease, active bleeding within 3 months, congenital renal disease (e.g., polycystic kidney disease) or disorder, with head injury or meningitis 3 months prior to dosing, in the opinion of the investigator or any uncontrolled medical illness which in the opinion of the investigator would jeopardize the safety of the subject, interfere with study assessments, or impact the validity of the study results.
* Known history of or positive screening result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCVAb).
* Subject has a positive test result for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) viral RNA test on Day -1.
* Subject who has a known, or suspected allergy, or sensitivity to polymyxins (colistin, polymyxin B) antibiotics in the opinion of the investigator.
* Subject with current evidence or history of malignancy in the 1 year prior to Day -1.
* Subject who has received polymyxins (colistin, polymyxin B) treatment within 28 days prior to Day -1.
* Use of prohibited medications of this study within 28 days (or 5 half-lives, if longer) prior to Day -1.
* Subjects with a QT interval corrected using Fridericia's formula (QTcF) prolongation over 500 milliseconds or history of prolonged QT syndrome at screening.
* Subject who used other investigational medicine within 28 days prior to the screening visit or plan to use other investigational medicine during the study period.
* Donation of blood within 56 days or plasma within 14 days prior to the screening visit or plan to donate during the entire study period.
* Blood transfusion within 14 days prior to the screening visit or necessary for regular blood transfusion within 3 months prior to the screening visit.
* Reports of a history of substance or alcohol abuse within 1 year prior to the screening visit.
* Female subject who is currently pregnant or breastfeeding or plans to be pregnant during the study period.
* Unstable or new medical conditions in the 3 months prior to screening.
* Any condition determined by the investigator to be unsuitable for subject enrollment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Cmax | Baseline,48hours
  Cmax: Maximum observed plasma concentration
AUC0-last | Baseline,48hours
  AUC0-last: Area under the plasma concentration vs time curve from time 0 to the last measurable concentration
AUC0-inf | Baseline,48hours
  AUC0-inf: Area under the plasma concentration vs time curve from time 0 extrapolated to infinity
CL | Baseline,48hours
  CL: Clearance, calculated as Dose/AUC0-inf

CONTACTS AND LOCATIONS:
Overall Officials: Fang, Principal Investigator — Shin Kong Memorial Wu Ho-Su Hospital
Locations (1):
- Shin Kong Memorial Wu Ho-Su Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No individual participant data(IPD) sharing plan